CLINICAL TRIAL: NCT02825823
Title: The Effects of Exogenous Ketones on Exercise Performance in Young Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H1601260
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Exercise; Ketones; Dietary Supplements
MeSH Terms: conditions — Motor Activity; Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketone Salts (Experimental): Acute dose of beta-hydroxybutyrate potassium/sodium salt (0.2g beta-hydroxybutyrate/kg, 0.01g Potassium/kg, 0.01g Sodium/kg with 1 g Steviol Glycoside and 30 ml of lemon juice per dose)
  Interventions: Dietary Supplement: Ketone Salt
- Placebo (Placebo Comparator): Acute dose of taste-matched placebo (0.01g Potassium/kg, 0.01g Sodium/kg with 1 g Steviol Glycoside and 30 ml of lemon juice per dose)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone Salt
  Arms: Ketone Salts
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The ketone body beta-hydroxybutyrate is produced during prolonged fasting or exercise and can be used as an alternative fuel source. Exogenous beta-hydroxybutyrate, in the form of a ketone salt, is proposed to have ergogenic potential for high-intensity exercise performance but this has not been adequately studied. The purpose of this study is to determine whether supplementing with an acute dose of ketone salts can alter fuel use during exercise and improve exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-40
* Ability to understand and communicate in English to answer questionnaires and interact with the research assistant
* Physically active (defined by engaging in moderate-to-vigorous exercise at least 3 times per week, determined via validated questionnaire)

Exclusion Criteria:

* Diagnosed with diabetes or any other medical conditions that could affect metabolism.
* Diagnosed with heart disease or taking anti-hypertensive medications.
* Competitive endurance athlete (self-identified as engaged in specific endurance training in triathlon, cycling, or distance running and competing in races or competition)
* Recent (last 3 months) or current consumption of a low-carbohydrate ketogenic diet
* Current consumption of ketone supplements
* Any other contraindication to vigorous exercise (identified via physical activity readiness questionnaire [PAR-Q])

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Respiratory Exchange Ratio (RER) during cycling exercise | 0-18 minutes
  The RER during 18 minutes of steady-state exercise

SECONDARY OUTCOMES:
10 km Cycling Time Trial Performance | Following 18 minutes of steady-state exercise
  10 km time trial performed on a stationary bicycle following 18 minutes of steady-state exercise

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada